CLINICAL TRIAL: NCT03840447
Title: Analysis of the Efficiency of a Chronic Disease Self-Management Programme in Population With Socioeconomic Vulnerability in Five European Countries
Brief Title: Analysis of the Efficiency of a Chronic Disease Self-Management Programme in a Vulnerable Population in Five European Countries
Acronym: EFFICHRONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Ente Ospedaliero Ospedali Galliera (Other); Erasmus Medical Center (Other); Asturias Public Health Service (SESPA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL19_0005; 2018-A01054-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-26; First posted 2019-02-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-01

CONDITIONS: Chronic Disease
Keywords: Chronic Disease; Prevention and control; Patient Education as Topic; Health Services/utilization; Program Evaluation; Cost-Benefit Analysis; Self-Efficacy; Disease Management; Health Status; Outcome Assessment (Health Care); Self Care; Socioeconomic Factors; Poverty Areas; Chronic Disease Self-Management Programme
MeSH Terms: conditions — Chronic Disease; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic Disease Self-Management programme (Experimental)
  Interventions: Behavioral: Chronic Disease Self-Management programme

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management programme — The primary aim of the intervention is to achieve greater self-management of the chronic condition by changing the role of the passive citizen to empowerment in self-confidence and self-reliance. The intervention consists of a series of 6 workshops (with 7 to 8 activities), 2.5 hours each, which are held once a week for 6 weeks. One professional and one peer will volunteer together to lead a series of workshops. To this end, professionals and peers will be recruited and trained in the CDSMP principles.
  Over 6 workshops, citizens set realistic health goals, learn to self-manage pain and discomfort, to self-manage their diet, self-manage physical activity, mood and the way the disease influences their personal relationships. The intervention is designed to actively involve citizens.

SUMMARY:
According to the World Health Organization (WHO), it is estimated that around 35% of women and 29% of men are affected by chronic conditions and this percentage is clearly influenced by specific risk factors, such as lifestyle indicators. The high prevalence of chronic conditions put a large burden on national budgets. The healthcare costs of chronic conditions reach 6.8% of GDP in some European countries. The economic factors are also conditioning the individuals' lifestyles, including their concerns about health and self-care as a part of their way of life. the most educated patients suffering from a chronic disorder have often better skills to manage their conditions and therefore, show better health indicators than those less educated or with lowest socioeconomic status. In addition, the former are normally more interested in participating in community-based interventions, training programmes and research actions. Thus, the impact of interventions targeted to increase self-management skills and improve health condition of individuals with chronic diseases could be extremely higher in those individuals with education and socioeconomic vulnerability traits. Several health education programs have shown positive effects in the self-management of chronic disease. The Chronic Disease Self-Management Programme is a program based on empowering people with chronic diseases to manage and control their disease. This program has been used in several countries over the past twenty years and its effectiveness has been widely demonstrated. However, this programme has not been specifically offered to people in situations of socio-economic vulnerability. The implementation of the EFFICHRONIC project, in five European countries with different health systems and socio-economic contexts, will validate the effectiveness of this program with vulnerable people with chronic diseases. Indeed, the investigators believe that the benefit of interventions aimed at increasing self-management skills and improving the health status of people with chronic diseases could be greater for people with socio-economic vulnerability characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Person older than 18 years of age who has one of the following condition:
2. Situation 1: Isolated Caregivers

   • Caregiver: a person that takes care of someone with an illness. The caregiver may be a spouse or partner, sibling, adult child, other family member or friend of someone with a chronic illness. Caregivers might be primary or secondary caregivers and live with or separate from the person receiving care. Caregivers don´t have to suffer from a chronic disease, but they must have a vulnerability condition defined as at least one of the following criteria:
   * without support network or
   * without means of transport or limited access to it (without private car and without public transport near to the place of residence (more than 1 km from the house)) or
   * digital isolation: without wifi or internet
3. Situation 2: Vulnerable people with a chronic disease

   * A chronic disease (self-reported or clinically evaluated by medical staff) according to the International Classification of Primary Care (ICPC-2): a chronic pathology with code between 70 and 99 registered in one of the 17 chapters (see Annex)
   * Chronic disease that has more than six months of evolution.
   * Vulnerability condition, such as:

     * Elderly people (older than 65 years of age) living alone or living in a nursing home and being in a situation of social or family isolation
     * Ethnic minorities (Travellers - Gens du Voyage) on a low income*
     * Legal immigrants, refugees and asylum-seekers on a low income*. For the asylum-seekers the domicile must be known for at least 6 months
     * Other vulnerable persons on a low income* even if not included in the previous target groups.

       * Low income: below the poverty line at 60 % of median standard of living for the year 2015 (see in the Annex, INSEE Première, 2017). We consider below the poverty line at 60 % the persons that are entitled to have: Revenu de Solidarité Active -RSA, Couverture Maladie Universelle Complémentaire - CMU-C, or Allocation Adulte Handicapé - AAH, or Allocation pour Demandeur d'Asile - ADA or Allocation de solidarité aux personnes âgées-ASPA. The persons that are entitled to have the Pension d'invalidité are included regardless their income. For all the others types of social allowance, the revenue should be below the poverty line at 60 % of median standard of living for the year 2015 (see in the Annex, INSEE Première, 2017).
4. Illiterate individuals older than 18 years of age who are in situation 1 or 2 might be included

Exclusion criteria:

1. - Person who could not commit to a 6-months follow-up regardless of the reason
2. Person living a period of crisis (domestic violence, refugees without a stable environment, eviction, etc.).
3. Basic housing needs not met (homeless or roofless).
4. Diagnosed with severe mental health problems (DSM V) (e.g. psychosis…) with distorted perception of reality and/or inability to function in a group.
5. Cognitive decline (e.g. Alzheimer´s), identified as a score from 0 to 42 on the "Test Your Memory" test.
6. Active addictive disorders (drugs, alcohol). If addiction took place in the past but at the time of inclusion the addiction is over, the person may be included
7. People without an adequate knowledge of the language of the country of residence.
8. Prisoners or subjects who are involuntary incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of a 6-weeks self-management program on the quality of life by SF-12 between baseline and 6 months | 6 months
  12-Item Short Form Health Survey (SF-12) has two components: physical composite scores (PCS) and mental composite scores (MCS). These two components measure eight concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems and mental health (psychological distress and psychological wellbeing). PCS and MCS are computed using the scores of twelve questions and the sum of PCS and MCS range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.

SECONDARY OUTCOMES:
Evaluation of the health status between baseline and 6 months | 6 months
  Evaluate the change in the health status change in score for : EQ-5D-5L questionnaire. EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The subject is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the subject's health state. The EQ VAS records the subject's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' (score 100) and 'The worst health you can imagine' (score 0). The VAS can be used as a quantitative measure of health outcome that reflect the subject's own judgement.
Evaluation of the wellbeing between baseline and 6 months | 6 months
  Evaluate the change in sleep, fatigue with standard 10 cm horizontal Visual Analogue Scales (VAS) anchored by no pain/fatigue and pain/fatigue as bad as it could be. Scores range between 0 and 10, with higher scores representing greater pain and fatigue. Shortness of breath was also measured with a standard 10 cm horizontal VAS (range 0-10) anchored by not at all and almost totally
Evaluation of the heatlhy behaviour between baseline and 6 months | 6 months
  Evaluate the 6-months change in physical exercise using exercise behaviours(scales which is designed for use in evaluations of the CDSMC (Lorig et al., 1999). Exercise was assessed in terms of duration (minutes per week) of exercises performed (e.g. stretching, strengthening, bicycling, swimming, etc.)) and IPAQ comprises a set of 5 activity domains: job-related physical activity, transportation physical activity, housework, house maintenance, and caring for family, recreation, sport, and leisure-time physical activity and time spent sitting. For this evaluation, the investigator assess only the time spent sitting domain, asking the duration (hours and minutes per day) of time spend sitting on a weekday and on a weekend. The value is average for the previous 4 weeks.
Evaluation of the communication with physician between baseline and 6 month | 6 months
  Communication with physician is assessed using three-item scales, with each item rated on a five-point scale (0-5) anchored by never and always. Scores for each scale are summed to produce total scores of 0-15, with higher scores indicating improved communication with physician.
Evaluation of the self-efficacy (confidence in ability to deal with health problems) between baseline and 6 month | 6 months
  Self-management is assessed using a self-efficacy -items scales on managing chronic disease. It covers several domains that are common across many chronic diseases: symptom control, role function, emotional functioning and communicating with physicians. Each item is scored from 1 (not at all confident) to 10 (totally confident). Scores are summed across the six items (range 5-60), with higher scores indicating greater self-efficacy.
Evaluate the cost-effectiveness of the program between baseline and 6 month | 6 months
  Cost-effectiveness is assessed using QALYs (quality-adjusted life years)obtained by the EQ-5D-5L descriptive system. It may be converted into a single index value. The index values are a major feature of the EQ-5D instrument, facilitating the calculation of (QALYs).
  HRQol (health-related quality of life) will be obtain using the SF-12. Four types of health care utilization were assessed: visits to GP, specialists and Accident and Emergency Units and number of nights spent in hospital. The questionnaire adopts a recall period of 6 months.
  Productivity Cost Questionnaire (PCQ) is a modified version of the 18 questions PCQ. The investigators collect 3 general questions: work status (number of hours per week of paid work and number of working days a week). Productivity losses measured in two separate modules: productivity losses of paid work due to absenteeism and presentism and productivity losses related to unpaid work. The questionnaire adopts a recall period of 4 weeks.
Evaluation of the adherence to treatment according to number of sessions performed | 6 months
  Evaluate the adherence to treatment between baseline and 6 month
Evaluate the medical error experience between baseline and 6 month | 6 months
  Medical error is assessed using three questions: 1 - the capacity of the healthcare provider to explain things, 2 - if the responder has experienced a medical error and 3- the seriousness of this error.
Evaluate the critical thinking between baseline and 6 month | 6 months
  Critical thinking and improved selection of information is assessed by two items of the Consortium for the European Health Literacy Survey on accessing Healthcare information and understanding. Each item is rated on a five-point scale (1-4) anchored by very difficult and very easy while the score "5" corresponds to "I don't know". Scores for each scale are summed to produce total scores of 2-10, with a scores of 8 indicating the higher health literacy.
Evaluate the improved selection of information between baseline and 6 month | 6 months
  Critical thinking and improved selection of information is assessed by two items of the Consortium for the European Health Literacy Survey on accessing Healthcare information and understanding. Each item is rated on a five-point scale (1-4) anchored by very difficult and very easy while the score "5" corresponds to "I don't know". Scores for each scale are summed to produce total scores of 2-10, with a scores of 8 indicating the higher health literacy.
Evaluate the impact of the program CDSMP at 6 months | 6 months
  Evaluation of the program is estimated by the improvement in the self-management techniques which is assessed by two items that scores from 0 (strongly disagree) to 4 (strongly agree) with higher score indicating greater ability in the self-management techniques and in the improvement in the decision making, interpersonal communication, confidence National Health System assessed by four items that scores from 0 (not at all) to 4 (extremely) with higher score indicating greater ability in decision making, interpersonal communication, confidence National Health System The satisfaction survey of the CDSMP is assessed at 6-months by a scored from 1 (not at all satisfied) to 10 (totally satisfied) with higher scores indicating greater satisfaction. At 6 weeks a survey to evaluate the satisfaction in the organisation of the program by five items (welcoming, clarity of the program, documents provided, activities done and location) will be given to the participants, as requested by the ARS.
Description of the characteristics of population included in the project | 6 months
  Description of the characteristics of population included in the project according to a self-administrated multidimensional prognostic indices which includes social determinants (SELFY-MPI)
Assess the influence of the type of help during the baseline visit and at 6 months visit | 6 months
  Influence of the help during the filling out process of questionnaires is assessed by three items: reason why the external help is required, who is helping the participants to fill out the questionnaire and school level of the participant.
Evaluation of the wellbeing between baseline and 6 months | 6 months
  Evaluate the change in depression with questionnaire PHQ-8. It consists of eight of the nine criteria on which the DSM-IV diagnosis of depressive disorders is based: depressed mood or irritable, decreased interest or pleasure, significant weight change (5%) or change in appetite, change in sleep, change in activity, fatigue or loss of energy, guilt/worthlessness and concentration. The subject is asked to indicate how often she/he had this problem over the last two week. Each criteria scores as "0" (not at all), "1" (several days), "2" (more than half of days) or "3" (nearly every day). Score is the sum of the 8 items. A score of 10 or greater is considered major depression, 20 or more is severe major depression
Evaluation of the heatlhy behaviour between baseline and 6 months | 6 months
  Evaluate the 6-months change in healthy eating by three items: eating breakfast, eating fruits and vegetables on a week. Because it is difficult to get good self-report data about nutrition, we use these three questions as surrogates for more generalized data about eating habits.
Evaluation of the heatlhy behaviour between baseline and 6 months | 6 months
  Evaluate the 6-months change in alcohol consumption is assessed by one domain of the Alcohol use disorders test: Hazardous alcohol use. The item that is here considered is the frequency of drinking. The score goes from 0 (no consummation of drinks containing alcohol) to 4 (4 or more drinks containing alcohol in a week).
Evaluation of the heatlhy behaviour between baseline and 6 months | 6 months
  Evaluate the 6-months change in smoking by a question with a yes/no answer

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology department, Montpellier, France

IPD SHARING:
Plan to Share IPD: No